CLINICAL TRIAL: NCT02213575
Title: Study 3: Effect of Minocycline Treatment on Drug-Resistant Hypertensive Patients
Brief Title: Study 3: Minocycline Decreases Microglia Activation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201500594 -N; RO1HL3361028 (Other: National Heart, Lung and Blood Institute (NHLBI)); 2013-00102 Study 3 (Other: Univeristy of Florida); R01HL132448 (NIH)
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Results first posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2023-05

CONDITIONS: Hypertension
Keywords: Resistent Hypertension
MeSH Terms: conditions — Hypertension | interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Minocycline Treatment Group (Experimental): Participants with neurogenic treatment-resistant hypertension who meet inclusion/exclusion criteria will receive minocycline at a dose determined to be most effective in lowering blood pressure (based on results from Study 1).
  Participants will undergo brain imaging with MRI and PET at baseline and 26 weeks.
  Intervention:
  Drug: Minocycline Dose: 50, 100, or 200 mg/day (based on optimal BP-lowering dose from Study 1) Frequency: Administered orally twice daily (BID) Duration: 26 weeks
  Interventions: Drug: Minocycline
- Control (No Intervention): Patients without a diagnosis of neurogenic (treatment-resistant) Hypertension and have not been treated with minocycline will be recruited. These participants will undergo one-time brain imaging visit (MRI and PET)

INTERVENTIONS:
Drug: Minocycline — Subjects will receive the dose of Minocycline determined to best lower BP and will undergo baseline and 26 week follow-up MRI and PET scans for changes in the paraventricular nucleus.
  Arms: Minocycline Treatment Group

SUMMARY:
This study is a mechanistic study that will enroll 9 subjects who are participating in NCT02133872 (which is designed to evaluate minocycline to test the hypothesis that minocycline treatment would produce antihypertensive effects in drug-resistant neurogenic hypertensive individuals) to test whether the antihypertensive effect of minocycline is associated with a decrease in activated microglia in central nervous system autonomic regions as evidenced by changes in PET and MRI imaging.

DETAILED DESCRIPTION:
This study (Study 3) will recruit 9 subjects from NCT02133872 (Study1) who will agree to undergo additional autonomic testing and imaging studies at baseline and after 6 months of study treatment. Specialized imaging of the brain using magnetic resonance imaging (MRI) and positron emission tomography (PET) scanning will be conducted at the Montreal Neurological Institute, in Montreal Canada.

For this study (Study 3) we include participants being enrolled Study 1 and/or participants who have completed participation in Study 1 and have not taken minocycline for 2 months will be approached to enroll in Study 3.

ELIGIBILITY:
Inclusion Criteria for Minocycline Subjects:

* Subjects participating in Study 1 will be eligible to participate.
* (For Study 3 Participants only) Willing to travel to Montreal, Canada for specialized imaging of the participant's brain using magnetic resonance imaging (MRI), positron emission tomography (PET) scanning, Autonomic Nervous System Testing and blood drawing- if participant qualifies

Exclusion Criteria for Minocycline Subjects:

-Female participants with positive pregnancy test.

Inclusion Criteria for Controls:

* No diagnosis of neurogenic (treatment-resistant) hypertension.
* Not treated with minocycline.
* Willing to travel to Montreal, Canada for brain imaging and testing.
* Able to provide informed consent.

Exclusion Criteria for Controls:

-Female participants with positive pregnancy test.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-03-05 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Pepine, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health Cardiovascular Clinic, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Minocycline Treatment Group: Participants with neurogenic treatment-resistant hypertension who meet inclusion/exclusion criteria will receive minocycline at a dose determined to be most effective in lowering blood pressure (based on results from Study 1).
  Participants will undergo brain imaging with MRI and PET at baseline and 26 weeks.
  Intervention:
  Drug: Minocycline Dose: 50, 100, or 200 mg/day (based on optimal BP-lowering dose from Study 1) Frequency: Administered orally twice daily (BID) Duration: 26 weeks
  Minocycline: Subjects will receive the dose of Minocycline determined to best lower BP and will undergo baseline and 26 week follow-up MRI and PET scans for changes in the paraventricular nucleus.
Period: Overall Study
Arm/Group | Minocycline Treatment Group | Control
Started | 5 | 0
Completed | 5 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Controls could not be recruited for this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Minocycline Treatment Group | Control | Total
Number analyzed (Participants) | 5 | 0 | 5
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.20 (3.70) |  | 69.20 (3.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 |  | 3
  Male | 2 |  | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 5 |  | 5
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 |  | 5

OUTCOME MEASURES:

1. Primary Outcome: PET Changes in the Paraventricular Nucleus From Baseline to 26 Weeks.
Description: This outcome represents the change in PET signal intensity in the bilateral paraventricular nucleus before and after minocycline treatment. PET imaging was performed using the radiotracer [¹¹C]PBR28, which binds to the Translocator Protein (TSPO), a marker of activated microglia and neuroinflammation. To ensure accurate anatomical localization, each participant's PET scan was co-registered with a high-resolution T1-weighted MRI. Regions of interest (ROIs) were manually drawn on the MRI and applied to the PET images to extract PET signal from the same brain structures. The signal was quantified as non-displaceable binding potential (BP_ND). The change in signal is calculated as the average change in BP_ND at baseline minus the average change in BP_ND after treatment. A positive value indicates that the PET signal decreased following treatment, reflecting a reduction in microglial activation and suggesting a favorable anti-inflammatory response to minocycline.
Time Frame: Change in Baseline to 26 weeks
Population: One subject was identified as a slow metabolizer of [¹¹C]PBR28 and therefore their data could not be used.
Measure: Mean (Standard Deviation); unit: Binding Potential (non-displaceable)
Arm/Group | Minocycline Treatment Group | Control
Number analyzed (Participants) | 4 | 0
Binding Potential (non-displaceable) | 0.0350 (0.0292) |

ADVERSE EVENTS:
Time Frame: 26 weeks
Description: No controls were recruited for this study therefore number of participants at risk for Serious Adverse Events, All-Cause Mortality and Other (Not Including Serious) Adverse Events is zero
Arm/Group | Minocycline Treatment Group | Control
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/0
Other Adverse Events (participants affected / at risk) | 0/5 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/75/NCT02213575/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/75/NCT02213575/ICF_001.pdf